CLINICAL TRIAL: NCT03911713
Title: A Phase 2, Randomized, Double-blind Study to Evaluate the Efficacy and Safety of VX-561 in Subjects Aged 18 Years and Older With Cystic Fibrosis
Brief Title: A Phase 2 Study to Evaluate Efficacy and Safety of VX-561 in Subjects Aged 18 Years and Older With Cystic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX18-561-101; 2018-003970-28 (EudraCT Number)
Record Dates: First submitted 2019-04-09; First posted 2019-04-11 (Actual); Results first posted 2022-01-25 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2021-12

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — ivacaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Ivacaftor (Active Comparator): Participants received IVA 150 milligrams (mg) orally every 12 hours (q12h) in the treatment period for 12 weeks.
  Interventions: Drug: IVA; Drug: Placebo
- VX-561: 25 mg (Experimental): Participants received VX-561 25 mg orally daily (qd) in the treatment period for 12 weeks.
  Interventions: Drug: VX-561; Drug: Placebo
- VX-561: 50 mg (Experimental): Participants received VX-561 50 mg orally qd in the treatment period for 12 weeks.
  Interventions: Drug: VX-561; Drug: Placebo
- VX-561: 150 mg (Experimental): Participants received VX-561 150 mg orally qd in the treatment period for 12 weeks.
  Interventions: Drug: VX-561; Drug: Placebo
- VX-561: 250 mg (Experimental): Participants received VX-561 250 mg orally qd in the treatment period for 12 weeks.
  Interventions: Drug: VX-561; Drug: Placebo

INTERVENTIONS:
Drug: VX-561 — VX-561 tablets for oral administration.
  Other Names: CTP-656; Deutivacaftor (D-IVA)
  Arms: VX-561: 150 mg; VX-561: 25 mg; VX-561: 250 mg; VX-561: 50 mg
Drug: IVA — 150-mg film-coated tablet for oral administration.
  Other Names: VX-770; Ivacaftor
  Arms: Ivacaftor
Drug: Placebo — Placebo matched to IVA.
  Arms: VX-561: 150 mg; VX-561: 25 mg; VX-561: 250 mg; VX-561: 50 mg
Drug: Placebo — Placebos matched to VX-561.
  Arms: Ivacaftor

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, pharmacodynamic (PD) and pharmacokinetic (PK) effect of VX-561.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have 1 of the following 9 CFTR mutations on at least 1 allele: G551D, G178R, S549N, S549R, G551S, G1244E, S1251N, S1255P, or G1349D
* On ivacaftor therapy
* FEV1 value ≥40% and ≤100% of predicted mean for age, sex, and height

Key Exclusion Criteria:

* History of clinically significant cirrhosis with or without portal hypertension
* History of solid organ or hematological transplantation
* Lung infection with organisms associated with a more rapid decline in pulmonary status

Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-08-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (48):
- United States (30):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Banner University of Arizona Medical Center, Tucson, Arizona
  - Miller Children's Hospital / Long Beach Memorial, Long Beach, California
  - UCSF Gateway Medical Center, San Francisco, California
  - National Jewish Health, Denver, Colorado
  - University of Miami Miller School of Medicine, Miami, Florida
  - Central Florida Pulmonary Group, PA, Orlando, Florida
  - Indiana University, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital Cystic Fibrosis Center Clinical Research Center, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Michigan Medicine, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Washington University School of Medicine / St. Louis Children's Hospital, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Columbia University Medical Center, New York, New York
  - University of North Carolina Hospitals, Chapel Hill, North Carolina
  - UC Health Holmes, Cincinnati, Ohio
  - ProMedica Toledo Hospital/Toledo Children's Hospital/Pediatric Pulmonary & Cystic Fibrosis Center, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Dell Children's Medical Group, Austin, Texas
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Utah / Primary Children's Medical Center, Salt Lake City, Utah
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Australia (4):
  - The Prince Charles Hospital, Chermside
  - Alfred Hospital, Melbourne, VIC
  - Mater Adult Hospital, South Brisbane
  - Westmead Hospital, Westmead
- Universitair Ziekenhuis Gent, Ghent, Belgium
- Germany (5):
  - Friedrich-Alexander University of Erlangen-Nuremberg, University Children's Hospital, Erlangen
  - Ruhrlandklinik Westdeutsches Lungenzentrum am Klinikum Essen, Essen
  - Universitätsklinikum Halle (Saale) / Universitätsklinik und Poliklinik für Innere Medizin, Schwerpunkt Pneumologie, Halle
  - Pneumologisches Studienzentrum Muenchen-West, München
  - University Hospital Wuerzburg, Würzburg
- Ireland (4):
  - Beaumont Hospital, Dublin
  - Cork University Hospital, Dublin
  - St. Vincent's University Hospital, Dublin
  - University Hospital Limerick (Adults), Limerick
- UMC St. Radboud, Nijmegen, Netherlands
- United Kingdom (3):
  - Clinical Research Facility, Queen Elizabeth University Hospital, Glasgow
  - St. James University Hospital, Leeds
  - Liverpool Heart and Chest Hospital, Liverpool

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing

REFERENCES:
- [Derived] Uluer AZ, MacGregor G, Azevedo P, Indihar V, Keating C, Mall MA, McKone EF, Ramsey BW, Rowe SM, Rubenstein RC, Taylor-Cousar JL, Tullis E, Yonker LM, Chu C, Lam AP, Nair N, Sosnay PR, Tian S, Van Goor F, Viswanathan L, Waltz D, Wang LT, Xi Y, Billings J, Horsley A; VX18-121-101; VX18-561-101 Study Groups. Safety and efficacy of vanzacaftor-tezacaftor-deutivacaftor in adults with cystic fibrosis: randomised, double-blind, controlled, phase 2 trials. Lancet Respir Med. 2023 Jun;11(6):550-562. doi: 10.1016/S2213-2600(22)00504-5. Epub 2023 Feb 23. PMID 36842446

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted in cystic fibrosis (CF) participants aged 18 years or older who have a gating mutation and were previously taking stable dose of ivacaftor (IVA).
Groups:
- VX-561: 25 mg: Participants received VX-561 25 mg orally once daily (qd) in the treatment period for 12 weeks.
Period: Overall Study
Arm/Group | Ivacaftor | VX-561: 25 mg | VX-561: 50 mg | VX-561: 150 mg | VX-561: 250 mg
Started | 12 | 6 | 11 | 24 | 24
Full Analysis Set (Received at least 1 dose of study drug in treatment period.) | 11 | 6 | 11 | 23 | 24
Completed | 11 | 4 | 11 | 22 | 24
Not Completed | 1 | 2 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 1 | 0
Not completed — Randomized, Never Dosed | 1 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ivacaftor: Participants received IVA 150 mg orally q12h in the treatment period for 12 weeks.
- VX-561: 25 mg: Participants received VX-561 25 mg orally qd in the treatment period for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Ivacaftor | VX-561: 25 mg | VX-561: 50 mg | VX-561: 150 mg | VX-561: 250 mg | Total
Number analyzed (Participants) | 11 | 6 | 11 | 23 | 24 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.3 (11.7) | 33.0 (10.6) | 27.8 (9.0) | 32.5 (8.5) | 37.4 (11.4) | 33.5 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 3 | 8 | 9 | 26
  Male | 7 | 4 | 8 | 15 | 15 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 11 | 6 | 10 | 22 | 24 | 73
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 10 | 6 | 11 | 23 | 24 | 74
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) [Mean (Standard Deviation); unit: percentage points] — FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
  percentage points | 74.0 (21.2) | 63.6 (22.4) | 66.8 (17.4) | 72.6 (17.3) | 73.9 (17.0) | 71.6 (18.0)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1)
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: From Baseline at Week 12
Population: Full analysis set (FAS) included all randomized participants who have intended CF transmembrane conductance regulator gene (CFTR) genotype and received at least 1 dose of study drug in treatment period. VX-561:25 mg and VX-561:50 mg arms were discontinued at sponsor's discretion and it was specified in statistical plan that data will be reported for only IVA, VX-561:150 mg and VX-561:250 mg arms for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage points
Arm/Group | Ivacaftor | VX-561: 150 mg | VX-561: 250 mg
Number analyzed (Participants) | 11 | 23 | 24
percentage points | -0.8 [-6.2 to 4.7] | 3.1 [-0.8 to 7.0] | 2.7 [-1.0 to 6.5]

2. Secondary Outcome: Absolute Change in Sweat Chloride (SwCl)
Description: Sweat samples were collected using an approved collection device.
Time Frame: From Baseline at Week 12
Population: FAS. VX-561:25 mg and VX-561:50 mg arms were discontinued at sponsor's discretion and it was specified in statistical plan that data will be reported for only IVA, VX-561:150 mg and VX-561:250 mg arms for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimole per liter (mmol/L)
Arm/Group | Ivacaftor | VX-561: 150 mg | VX-561: 250 mg
Number analyzed (Participants) | 11 | 23 | 24
millimole per liter (mmol/L) | 0.9 [-9.5 to 11.3] | 3.3 [-4.6 to 11.2] | -6.5 [-14.1 to 1.2]

3. Secondary Outcome: Observed Pre-Dose Concentration (Ctrough) of VX-561 and Its Metabolites (M1-VX-561 and M6-VX-561) and IVA and Its Metabolites (M1-IVA and M6-IVA)
Time Frame: At Week 4
Population: Pharmacokinetic (PK) set included all participants who received at least 1 dose of study drug and for whom the primary PK data were considered to be sufficient and interpretable. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "Number Analyzed" signifies those who were evaluable for the specific category.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Ivacaftor | VX-561: 25 mg | VX-561: 50 mg | VX-561: 150 mg | VX-561: 250 mg
Number analyzed (Participants) | 9 | 4 | 7 | 20 | 20
nanogram per milliliter (ng/mL)
  VX-561: Week 4: number analyzed (Participants) | 0 | 4 | 7 | 20 | 20
  VX-561: Week 4 |  | 26.1 (24.7) | 123 (61.6) | 458 (273) | 1100 (856)
  M1-VX-561: Week 4: number analyzed (Participants) | 0 | 4 | 7 | 20 | 20
  M1-VX-561: Week 4 |  | 18.1 (17.7) | 108 (58.6) | 378 (213) | 739 (407)
  M6-VX-561: Week 4: number analyzed (Participants) | 0 | 3 | 7 | 20 | 20
  M6-VX-561: Week 4 |  | NA (NA) — NA indicates that summary statistics were not reported as the number of observations below the limit of quantification was greater than 50% of the total number of observations at the specified time points. | 59.8 (34.0) | 211 (189) | 370 (233)
  IVA: Week 4: number analyzed (Participants) | 9 | 0 | 0 | 0 | 0
  IVA: Week 4 | 952 (766) |  |  |  |
  M1-IVA: Week 4: number analyzed (Participants) | 9 | 0 | 0 | 0 | 0
  M1-IVA: Week 4 | 1330 (774) |  |  |  |
  M6-IVA: Week 4: number analyzed (Participants) | 9 | 0 | 0 | 0 | 0
  M6-IVA: Week 4 | 662 (398) |  |  |  |

4. Secondary Outcome: Safety and Tolerability as Assessed by Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: Baseline up to Week 16
Population: Safety Set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Ivacaftor | VX-561: 25 mg | VX-561: 50 mg | VX-561: 150 mg | VX-561: 250 mg
Number analyzed (Participants) | 11 | 6 | 11 | 23 | 24
participants
  Participants with AEs | 8 | 4 | 8 | 21 | 23
  Participants with SAEs | 1 | 2 | 2 | 2 | 1

ADVERSE EVENTS:
Time Frame: Baseline up to Week 16
Arm/Group | Ivacaftor | VX-561: 25 mg | VX-561: 50 mg | VX-561: 150 mg | VX-561: 250 mg
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/6 | 0/11 | 0/23 | 0/24
Serious Adverse Events (participants affected / at risk) | 1/11 | 2/6 | 2/11 | 2/23 | 1/24
Other Adverse Events (participants affected / at risk) | 8/11 | 4/6 | 8/11 | 17/23 | 20/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ivacaftor (N=11) | VX-561: 25 mg (N=6) | VX-561: 50 mg (N=11) | VX-561: 150 mg (N=23) | VX-561: 250 mg (N=24)
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 1 | 1 | 2 | 2 | 1
Forced expiratory volume decreased (Investigations) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ivacaftor (N=11) | VX-561: 25 mg (N=6) | VX-561: 50 mg (N=11) | VX-561: 150 mg (N=23) | VX-561: 250 mg (N=24)
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Glaucoma (Eye disorders) | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Epididymitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 2 | 0 | 2 | 2 | 4
Nasopharyngitis (Infections and infestations) | 2 | 0 | 0 | 0 | 3
Oral candidiasis (Infections and infestations) | 1 | 1 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 2 | 1 | 1
Atypical mycobacterium test positive (Investigations) | 0 | 0 | 1 | 0 | 0
Bacterial test positive (Investigations) | 1 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 2 | 0 | 1
Blood glucose increased (Investigations) | 1 | 0 | 0 | 0 | 0
Coronavirus test positive (Investigations) | 1 | 0 | 0 | 0 | 0
Forced expiratory volume decreased (Investigations) | 0 | 1 | 1 | 0 | 0
Protein urine present (Investigations) | 1 | 0 | 0 | 0 | 0
Pulmonary function test decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Urine ketone body present (Investigations) | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 2 | 1
Sinus headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 6 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 1
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 2 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 4 | 0
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 1
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 4 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 4 | 3
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-10-03): https://cdn.clinicaltrials.gov/large-docs/13/NCT03911713/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-24): https://cdn.clinicaltrials.gov/large-docs/13/NCT03911713/SAP_001.pdf